CLINICAL TRIAL: NCT04022343
Title: A Phase 2 Study of Neoadjuvant Cabozantinib in Patients With Locally Advanced Non-Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Neoadjuvant Cabozantinib in Treating Patients With Locally Advanced Kidney Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Exelixis (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mehmet Bilen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00110583; NCI-2019-02253 (Other: NCI Clinical Trials Reporting Program); Winship4643-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Clear Cell Renal Cell Carcinoma; Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib) (Experimental): Patients receive cabozantinib orally once daily for 12 weeks in the absence of disease progression or unacceptable toxicity. The assigned starting dose for cabozantinib is 60 mg/day. Two dose reduction levels of cabozantinib are permitted
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Given PO
  Other Names: Cometriq; Cabometyx; BMS-907351; XL184; 1140909-48-3

SUMMARY:
This phase II clinical trial studies how well cabozantinib works in treating patients with kidney cancer before surgery. Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the objective response rate (complete and partial responses), following the administration of cabozantinib for 12 weeks in patients with locally advanced biopsy-proven non-metastatic clear cell renal cell carcinoma (ccRCC) prior to undergoing surgery.

SECONDARY OBJECTIVES:

I. To assess the safety, and tolerability of neoadjuvant cabozantinib.

II. To determine the clinical outcome (disease-free survival [DFS], overall survival [OS]) of patients with non-metastatic ccRCC who treated with neoadjuvant cabozantinib.

III. To evaluate the surgery related outcomes.

IV. To evaluate correlative studies, including biomarkers, quality of life, and frailty/sarcopenia assessment of patients with non-metastatic ccRCC who treated with neoadjuvant cabozantinib.

OUTLINE:

Patients receive cabozantinib orally (PO) once daily (QD) for 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal mass consistent with a clinical stage ≥ T3Nx or TanyN+ or deemed unresectable by surgeon.
* Renal cell carcinoma with clear cell component on pre-treatment biopsy of the primary tumor.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Patients must have adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

  * Absolute neutrophil count (ANC) ≥ 1500/mm³ (≥ 1.5 GI/L) without granulocyte colony-stimulating factor support.
  * White blood cell count ≥ 2500/mm³ (≥ 2.5 GI/L).
  * Platelets ≥ 100,000/mm³ (≥ 100 GI/L) without transfusion.
  * Hemoglobin ≥ 9 g/dL.
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). ALP ≤ 5 x ULN with documented bone metastases.
  * Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert's disease ≤ 3 x ULN).
  * Serum albumin ≥ 2.8 g/dl.
  * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft-Gault equation:

    * Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)
    * Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
  * Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol).
* No hormonal therapy, chemotherapy, immunotherapy, or any other systemic therapy for a malignancy, in the 5 years prior to current study enrollment.
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.
* Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.

Exclusion Criteria:

* Evidence of metastatic disease on pre-treatment imaging.
* The subject has received of any type of cytotoxic, biologic or other systemic anticancer therapy for kidney cancer.
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
* Known brain metastases or cranial epidural disease.
* Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel). Allowed anticoagulants are the following:

  * Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
  * Low-dose low molecular weight heparins (LMWH) are permitted.
  * Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* The subject has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test ≥ 1.3 × the laboratory ULN within 14 days before the first dose of study treatment.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 6 months before first dose.
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, active inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.
  * Clinically significant hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.
  * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
  * Other clinically significant disorders that would preclude safe study participation.

    * Serious non-healing wound/ulcer/bone fracture.
    * Uncompensated/symptomatic hypothyroidism.
    * Moderate to severe hepatic impairment (Child-Pugh B or C).
* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Prolongation of the QT corrected for HR using Fridericia's method (QTcF) interval defined as > 500 msec per electrocardiogram (ECG) within 28 days before first dose of study treatment. Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
* Pregnant or lactating females.
* Inability to swallow tablets.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy. Patients with Gleason 6 (3+3) prostate cancer with previous treatment or on active surveillance may also be allowed on protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2026-03-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Asim Bilen, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilen MA, Vo BT, Liu Y, Greenwald R, Davarpanah AH, McGuire D, Shiradkar R, Li L, Nazha B, Brown JT, Williams S, Session W, Russler G, Caulfield S, Joshi SS, Narayan VM, Filson CP, Ogan K, Kucuk O, Carthon BC, Del Balzo L, Cohen A, Boyanton A, Prokhnevska N, Cardenas MA, Sobierajska E, Jansen CS, Patil DH, Nicaise E, Osunkoya AO, Kissick H, Master VA. Neoadjuvant cabozantinib restores CD8+ T cells in patients with locally advanced non-metastatic clear cell renal cell carcinoma: a phase 2 trial. Res Sq [Preprint]. 2024 Aug 8:rs.3.rs-4849400. doi: 10.21203/rs.3.rs-4849400/v1. PMID 39149474

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cabozantinib)
Started | 22
Completed | 17
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabozantinib)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 57 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate will be evaluated using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) criteria. All tumor measurements must be recorded in centimeters.
  For target lesions, a complete response (CR) is defined as the disappearance of all target lesions. A partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: At 12 weeks after cabozantinib dose
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (cabozantinib)
Number analyzed (Participants) | 17
Participants
  Partial Response | 6
  Stable Disease | 11

2. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival will be defined as the interval between time of surgery and the first tumor recurrence or death. Patients will be censored at time of last follow-up. Disease-free survival will be estimated with the Kaplan-Meier method.
Time Frame: From time of surgery to first tumor recurrence or death, assessed up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (cabozantinib)
Number analyzed (Participants) | 17
percentage of participants
  12 month survival rate | 82.4 [54.7 to 93.9]
  24 month survival rate | 76.5 [48.8 to 90.4]

3. Secondary Outcome: Overall Survival (OS)
Description: For overall survival, death from any cause will be defined as the event. Patients will be censored at time of last follow-up. Overall survival will be estimated with the Kaplan-Meier method.
Time Frame: From time of surgery to death from any cause, assessed up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (cabozantinib)
Number analyzed (Participants) | 17
percentage of participants
  12 month survival rate | 94.1 [65 to 99.1]
  24 month survival rate | 88.2 [60.6 to 96.9]

4. Secondary Outcome: Quality of Life Assessment: Functional Assessment of Cancer Therapy-Kidney Specific Index-19 (FKSI-19) Questionnaire
Description: Quality of life will be studied using the Functional Assessment of Cancer Therapy-Kidney Specific Index-19 (FKSI-19) questionnaire. The questionnaire consists of 19 statements that patients answer on a 0-4 scale ("Not at all" to "Very much"). Per the instrument's official scoring guidelines, items are then reverse scored as needed and summed to create a final score ranging from 0-76, where 76 indicates the best quality of life and 0 indicates the worst.
Time Frame: Baseline and weeks 6 and 12 after treatment initiation
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment (cabozantinib)
Number analyzed (Participants) | 17
score on a scale
  Baseline | 60 [54.6 to 65.4]
  Week 6 | 48.6 [43.2 to 54.1]
  Week 12 | 48.5 [43.4 to 53.6]

5. Secondary Outcome: Quality of Life Assessment: Functional Assessment of Cancer Therapy-Kidney Specific Index-19 (FKSI-19) Questionnaire
Description: Quality of life will be studied using the Functional Assessment of Cancer Therapy-Kidney Specific Index-19 (FKSI-19) questionnaire. The questionnaire consists of 19 statements such as "I have a lack of energy" and "I have pain" which are answered on a scale of 0-4, with 0 being "Not at all" and 4 being "Very much." The scale is 0-76 (0 = worst QoL, 76 = best QoL).
Time Frame: Baseline and weeks 6 and 12 after treatment initiation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment (cabozantinib)
Number analyzed (Participants) | 17
score on a scale
  Baseline | 64 [55 to 67]
  Week 6 | 51 [38 to 55]
  Week 12 | 48 [43 to 57]

6. Secondary Outcome: Frailty Assessment
Description: Frailty assessment will be studied using the Fried Frailty score. Domains to be assessed include shrinking, weakness, exhaustion, low activity, and slow walking speed. Scored on a total scale of 0-25 (from 5 variables, each 0-5). 0 = not frail, 25 = most frail.
Time Frame: Baseline and weeks 6 and 12 after treatment initiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (cabozantinib)
Number analyzed (Participants) | 17
score on a scale
  Baseline | 1.18 (1.33)
  Week 6 | 1.82 (1.47)
  Week 12 | 2.06 (1.39)

7. Secondary Outcome: Sarcopenia Assessment
Description: Sarcopenia assessment will be done by using baseline and week 12 scans via SliceOmatic version 5.0 by TomoVision program. Cross-sectional skeletal muscle area (SMA) at the L3 vertebra will be segmented to calculate the Skeletal Muscle Index (SMI = SMA cm² / height m²). Sarcopenia is defined as an SMI at or below the 25th percentile of age- and sex-specific reference values from the Fintelmann et al. (2024) Framingham Heart Study cohort.
Time Frame: Baseline and week 12 after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (cabozantinib)
Number analyzed (Participants) | 16
Participants
  Participants with Sarcopenia (baseline) | 9
  Participants with Sarcopenia (week12) | 9

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Treatment (Cabozantinib)
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabozantinib) (N=17)
Vascular disorders - Other, specify (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Death (General disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabozantinib) (N=17)
Hot flashes (Vascular disorders) | 1
Creatinine increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Fever (General disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Fecal incontinence (Gastrointestinal disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Gait disturbance (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 4
Diarrhea (Gastrointestinal disorders) | 10
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Suicidal ideation (Psychiatric disorders) | 1
Investigations - Other, specify (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 3
Oral dysesthesia (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Papulopustular rash (Infections and infestations) | 2
Dizziness (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hemoglobin increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Gallbladder perforation (Hepatobiliary disorders) | 1
Depression (Psychiatric disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Hypotension (Vascular disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Paresthesia (Nervous system disorders) | 3
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 2
Edema limbs (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
GGT increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04022343/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT04022343/ICF_003.pdf